CLINICAL TRIAL: NCT02282202
Title: Evaluation of Oscillatory Positive Expiratory Pressure (oPEP) in Bronchiectasis and COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROB0038
Record Dates: First submitted 2014-10-24; First posted 2014-11-04 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchiectasis
Keywords: Sputum; Bronchiectasis; Chronic Obstructive Pulmonary Disease; Airway clearance therapy; Oscillatory Positive Expiratory Pressure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Off/on for 3 weeks followed by on/off for 3 weeks (Other): Subjects are randomized to either Oscillating Positive Expiratory Pressure device (Aerobika ®) or no device for three weeks, then crossover for the following three weeks.
  Interventions: Device: Oscillating Positive Expiratory Pressure (Aerobika ®)

INTERVENTIONS:
Device: Oscillating Positive Expiratory Pressure (Aerobika ®) — The oPEP system (Aerobika ®) combines positive expiratory pressure therapy and airway vibrations to help mobilize pulmonary secretions. oPEP therapy (Aerobika ®) enforces a resistance to exhalation at the mouth, while the airway vibration technology transmits movements upstream during exhalation so that airway walls may become free from mucous. Subjects will take home the device and use four times daily during the active part of the study.
  There is only one intervention for this study. Subjects are "on" treatment for three weeks and "off" for the alternate three weeks.
  Other Names: oPEP (Aerobika ®)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of four times daily Positive Expiratory Pressure (oPEP) (Aerobika ®) maneuvers over three weeks in individuals with bronchiectasis and chronic obstructive pulmonary disease (COPD) with chronic sputum production. The investigators hypothesize that four times daily positive expiratory pressure using the Aerobika ® will significantly improve dyspnea, movement of mucus, St. George's Respiratory Questionnaire (SGRQ) score, and six-minute walk distance (6MWD) after three weeks of four times daily administration.

DETAILED DESCRIPTION:
Cough and sputum production are common in Bronchiectasis and chronic obstructive pulmonary disease (COPD), both of which are associated with significant morbidity and other adverse clinical outcomes. Airway clearance techniques (ACTs) such as afforded by oscillatory Positive Expiratory Pressure (oPEP) (Aerobika ®) aim to remove sputum from the lungs, however evidence of their efficacy during stable disease is unclear.

The objective of this study is to evaluate the safety and efficacy of four times daily Positive Expiratory Pressure maneuvers over three weeks in individuals with bronchiectasis and COPD with chronic sputum production. The oPEP device (Aerobika ®) combines positive expiratory pressure therapy and airway vibrations to help mobilize pulmonary secretions. oPEP therapy enforces a resistance to exhalation at the mouth while the airway vibration technology transmits movements upstream during exhalation so that airway walls may become free from mucus. An adjustable dial allows users to adjust the frequency and the flow resistance based on their individual needs. Subjects will take a device home and use four times daily during the active part of the study. We hypothesize that daily oPEP use will significantly improve dyspnea, movement of mucus, SGRQ score, and 6MWD after three weeks of four times daily administration.

This is a randomized cross-over unblinded study in 30 subjects: ten with bronchiectasis and 20 with COPD (with chronic bronchitis and chronic mucus production identified). Five subjects from the Bronchiectasis group and ten from the COPD group will start with oPEP and use for three weeks. All subjects will crossover at Visit Two after three weeks of oPEP therapy or three weeks of no therapy. Each subject will visit the centre on three occasions: Baseline, Crossover Visit, and Final Visit for approximately one hour each and will perform: 1) spirometry and plethysmography, 2) 6MWT, and 3) health status evaluation using a self-administered SGRQ. Subjects will first provide written informed consent and will complete: 1) SGRQ after inhaling 2-4 puffs (200-400µg) of the short-acting bronchodilator (eg. Salbutamol), 2) plethysmography and spirometry 35 (±five minutes) post-salbutamol. Vital signs will be documented and subjects will rest for approximately 15 minutes before the six-minute walk test (6MWT) post-salbutamol. Subjects will be given an oPEP therapy system (Aerobika ®) to use at home, four times per day. Instruction and training on the use of the device will be given at the baseline visit. Subjects will be required to return the device upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 40-85 with either a clinical diagnosis of bronchiectasis or COPD with chronic bronchitis and chronic mucous production identified
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject is ambulatory and can perform the 6MWT
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* FEV1 >25% predicted -FVC > 25% predicted and >0.5L

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material. Capacity to consent will be determined by either Dr. McCormack at the time of the clinic visit or Sandra Blamires, the study coordinator.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in sputum production | weekly for six weeks
  Change in sputum production from subject self-reported questionnaires performed weekly

SECONDARY OUTCOMES:
Six Minute Walk Distance (6MWD) | Baseline, 3-weeks (cross-over), 6-weeks
Pulmonary function measurements | Baseline, 3-weeks (cross-over), 6-weeks
  Pulmonary function measurements include FEV1 (Forced expiratory volume in 1 second); FVC (forced vital capacity); FEV1/FVC ratio; TLC (total lung capacity); RV (residual volume); DLCO (Diffusing capacity of the lung)
St. George's Respiratory Questionnaire (SGRQ) | Baseline, 3-weeks (cross-over), 6-weeks
Dyspnea (Patient Evaluation Questionnaire) | Completed weekly for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario; David G McCormack, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- Robarts Research Insitute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Cochrane GM, Webber BA, Clarke SW. Effects of sputum on pulmonary function. Br Med J. 1977 Nov 5;2(6096):1181-3. doi: 10.1136/bmj.2.6096.1181. PMID 589074
- [Background] Ambrosino N, Callegari G, Galloni C, Brega S, Pinna G. Clinical evaluation of oscillating positive expiratory pressure for enhancing expectoration in diseases other than cystic fibrosis. Monaldi Arch Chest Dis. 1995 Aug;50(4):269-75. PMID 7550205
- [Background] Oberwaldner B, Evans JC, Zach MS. Forced expirations against a variable resistance: a new chest physiotherapy method in cystic fibrosis. Pediatr Pulmonol. 1986 Nov-Dec;2(6):358-67. doi: 10.1002/ppul.1950020608. PMID 3543830
- [Derived] Capaldi DPI, Guo F, Xing L, Parraga G. Pulmonary Ventilation Maps Generated with Free-breathing Proton MRI and a Deep Convolutional Neural Network. Radiology. 2021 Feb;298(2):427-438. doi: 10.1148/radiol.2020202861. Epub 2020 Dec 8. PMID 33289613
- [Derived] Svenningsen S, Paulin GA, Sheikh K, Guo F, Hasany A, Kirby M, Rezai RE, McCormack DG, Parraga G. Oscillatory Positive Expiratory Pressure in Chronic Obstructive Pulmonary Disease. COPD. 2016;13(1):66-74. doi: 10.3109/15412555.2015.1043523. Epub 2015 Oct 2. PMID 26430763